CLINICAL TRIAL: NCT02609100
Title: Video Capsule Endoscopy Versus Colonoscopy in Patients With Melena and Negative Upper Endoscopy: A Randomized Controlled Trial
Brief Title: Video Capsule Endoscopy Versus Colonoscopy in Patients With Melena and Negative Upper Endoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201507101
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Gastrointestinal Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Videotape Recording; Endoscopy; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Capsule Endoscopy (Active Comparator): Randomization arm one is to video capsule endoscopy (VCE) a non-invasive procedure in which a patient swallows a disposable 1.0 X 2.5 cm 'pill' containing a camera electronically linked to equipment outside the patient which records images as it passes from the esophagus through the entire tract and is excreted in feces. It images the small intestine in areas beyond the reach of upper GI endoscopy and the terminal ileum and is similarly beyond the reach of colonoscopy. Its greatest use is in identifying points of bleeding and ulcers.
  Interventions: Procedure: Video Capsule Endoscopy; Device: 1.0 X 2.5 cm 'pill' containing a camera
- Next Day Colonoscopy (Active Comparator): Randomization arm two is to colonoscopy, a test that allows the doctor to look at the inner lining of the large intestine (rectum and colon). He or she uses a thin, flexible tube called a colonoscope to look at the colon.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Video Capsule Endoscopy — Video Capsule Endoscopy allows for imaging of the small intestine between the distant duodeno-jejunal junction, which is beyond the reach of upper GI endoscopy and the terminal ileum and is similarly beyond the reach of colonoscopy. It is of greatest use in identifying points of bleeding and ulcers.
  Arms: Video Capsule Endoscopy
Procedure: Colonoscopy — The colonoscopy helps find ulcers, tumors, and areas of inflammation or bleeding in the large intestine.
  Arms: Next Day Colonoscopy
Device: 1.0 X 2.5 cm 'pill' containing a camera
  Arms: Video Capsule Endoscopy

SUMMARY:
Acute gastrointestinal bleeding is a common medical problem. When patients with gastrointestinal bleeding present with melena (dark, tarry stool) the blood loss is usually originating in the upper gastrointestinal tract (esophagus, stomach or duodenum) and first step in evaluating the patient is an upper endoscopy; which allows direct visualization of the esophagus, stomach and duodenum. However, the cause of bleeding is located in the small bowel or colon in 20-30% of patients who present with melena. Traditionally colonoscopy has been the next test preformed if upper endoscopy does not identify the cause of melena/ gastrointestinal bleeding, however less than 25% of patients who present with melena have bleeding originating in the colon, and the remainder of patients have bleeding originating in the small intestine, which can only be fully evaluated with video capsule endoscopy (a pill camera which is swallowed and takes pictures while it travels thought the small bowel and colon). Currently patients only undergo video capsule endoscopy if colonoscopy does not identify the cause of bleeding. The investigators are preforming a randomized study which seeks to determine if colonoscopy or video capsule endoscopy is a better way to identify the cause of gastrointestinal bleeding in patients who present with melena and have normal findings on upper endoscopy. To do this the investigators will enroll patients who present with melena prior to their upper endoscopy and if the cause of bleeding is not identified at that time patients will be randomized to video capsule endoscopy (with the capsule being placed into the small bowel during the upper endoscopy) or next day colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

• Inpatients >18 years of age presenting with lower gastrointestinal bleeding and have melenic stool

Exclusion Criteria:

* Unable to provide written informed consent
* A probable bleeding source is identified on upper endoscopy
* Pregnancy or lactation
* Swallowing Disorder
* Unable to tolerate sedation or anesthesia due to medical co-morbidities
* Uncorrected coagulopathy (platelet count <50,000, INR> 2, PTT> 2x upper limit of normal)
* Known or suspected gastrointestinal obstruction or stricture
* Cardiac pacemaker or other implanted electromedical device
* Contraindication to bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir M Kushnir, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Center for Advanced Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Video Capsule Endoscopy | Next Day Colonoscopy
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Video Capsule Endoscopy: Randomization arm one is to video capsule endoscopy (VCE) a non-invasive procedure in which a patient swallows a disposable 1.0 X 2.5 cm 'pill' containing a camera electronically linked to equipment outside the patient which records images as it passes from the esophagus through the entire tract and is excreted in feces. It images the small intestine in areas beyond the reach of upper GI endoscopy and the terminal ileum and is similarly beyond the reach of colonoscopy. Its greatest use is in identifying points of bleeding and ulcers.
  Video Capsule Endoscopy: Video Capsule Endoscopy allows for imaging of the small intestine between the distant duodeno-jejunal junction, which is beyond the reach of upper GI endoscopy and the terminal ileum and is similarly beyond the reach of colonoscopy. It is of greatest use in identifying points of bleeding and ulcers.
  1.0 X 2.5 cm 'pill' containing a camera
- Total: Total of all reporting groups
Arm/Group | Video Capsule Endoscopy | Next Day Colonoscopy | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] | 71.5 [71 to 72] | 79.5 [72 to 87] | 75.5 [71 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Findings Defined as Lesions Considered to Have a High Potential for Bleeding to Participants With no Significant Findings From Video Capsule Endoscopy
Description: Video Capsule Endoscopy identifies clinically significant lesions defined as lesions considered to have high potential for bleeding, such as a large ulceration, tumor or typical angiomata
Time Frame: Up to twenty four hours
Measure: Count of Participants; unit: Participants
Arm/Group | Video Capsule Endoscopy
Number analyzed (Participants) | 2
Participants | 1

2. Primary Outcome: Number of Participants With Clinically Significant Findings Defined as Lesions Considered to Have a High Potential for Bleeding to Participants With no Significant Findings From Colonoscopy
Description: Colonoscopy identifies clinically significant lesions defined as lesions considered to have high potential for bleeding, such as a large ulceration, tumor or typical angiomata
Time Frame: Up to one hour
Measure: Count of Participants; unit: Participants
Arm/Group | Next Day Colonoscopy
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Therapeutic Yield of Video Capsule Endoscopy
Description: Therapeutic yield of video capsule endoscopy is defined as the proportion of endoscopies leading to a therapeutic intervention.
Time Frame: Up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Video Capsule Endoscopy
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Therapeutic Yield of Colonoscopy
Description: Therapeutic yield of colonoscopy is defined as the proportion of endoscopies leading to a therapeutic intervention.
Time Frame: Up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Next Day Colonoscopy
Number analyzed (Participants) | 2
Participants | 0

5. Secondary Outcome: Number of Blood Units Transfused
Description: Number of blood units transfused measured in units of packed red blood cells
Time Frame: Up to 60 days
Measure: Mean (Full Range); unit: Units of blood
Arm/Group | Video Capsule Endoscopy | Next Day Colonoscopy
Number analyzed (Participants) | 2 | 2
Units of blood | 3 [2 to 4] | 0 [0 to 0]

6. Secondary Outcome: Number of Diagnostic Studies Performed for Evaluation of Gastrointestinal Bleeding
Description: Includes repeat endoscopies or imaging
Time Frame: Up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Video Capsule Endoscopy | Next Day Colonoscopy
Number analyzed (Participants) | 2 | 2
Participants | 2 | 1

7. Secondary Outcome: Duration of Hospital Stay
Description: The duration of hospital stay will be recorded in number of days
Time Frame: Up to 60 days
Measure: Mean (Full Range); unit: Days
Arm/Group | Video Capsule Endoscopy | Next Day Colonoscopy
Number analyzed (Participants) | 2 | 2
Days | 8 [6 to 10] | 14.5 [14 to 15]

8. Secondary Outcome: Procedure Related Adverse Events
Description: Adverse events related to the video capsule endoscopy and colonoscopy will be recorded
Time Frame: Up to 60 days
Measure: Number; unit: Adverse Events
Arm/Group | Video Capsule Endoscopy | Next Day Colonoscopy
Number analyzed (Participants) | 2 | 2
Adverse Events | 0 | 0

ADVERSE EVENTS:
Arm/Group | Video Capsule Endoscopy | Next Day Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Overall limit is that study was stopped and closed after only four successful enrollments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes